CLINICAL TRIAL: NCT03345836
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Induction Study of the Efficacy and Safety of Upadacitinib (ABT-494) in Subjects With Moderately to Severely Active Crohn's Disease Who Have Inadequately Responded to or Are Intolerant to Biologic Therapy
Brief Title: A Study of the Efficacy and Safety of Upadacitinib (ABT-494) in Participants With Moderately to Severely Active Crohn's Disease Who Have Inadequately Responded to or Are Intolerant to Biologic Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M14-431; 2017-001226-18 (EudraCT Number)
Record Dates: First submitted 2017-11-15; First posted 2017-11-17 (Actual); Results first posted 2022-08-15 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2022-07

CONDITIONS: Crohn's Disease
Keywords: Upadacitinib; Crohn's Disease; Efficacy; Safety
MeSH Terms: conditions — Crohn Disease | interventions — upadacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Part 1 (Double-blind): Placebo (Placebo Comparator): Participants received upadacitinib matching placebo tablets, orally, once daily (QD) for 12 weeks during the Double-blind (DB) Induction Period.
  Interventions: Drug: Matching Placebo for Upadacitinib
- Part 1 (Double-blind): Upadacitinib 45 mg (Experimental): Participants received upadacitinib 45 mg tablets, orally, QD for 12 weeks during the DB Induction Period.
  Interventions: Drug: Upadacitinib
- Part 2 (Open-label): Upadacitinib 45 mg (Experimental): Participants received upadacitinib 45 mg tablets, orally, QD for 12 weeks during the Open-label (OL) Induction Period.
  Interventions: Drug: Upadacitinib
- Part 3 (Extended Treatment DB): Upadacitinib 45 mg From Part 1 DB Placebo (Experimental): Participants received upadacitinib 45 mg tablets, orally, QD for 12 weeks (until Week 24) during the Extended Treatment (ET) Period. Participants who received placebo in Part 1 and did not achieve clinical response at Week 12 were included in this group.
  Interventions: Drug: Upadacitinib
- Part 3 (Extended Treatment DB): Upadacitinib 30 mg From Part 1 DB Upadacitinib 45 mg (Experimental): Participants received upadacitinib 30 mg tablets, orally, QD for 12 weeks (until Week 24) during the ET Period. Participants who received DB upadacitinib 45 mg in Part 1 and did not achieve clinical response at Week 12 were included in this group.
  Interventions: Drug: Upadacitinib
- Part 3 (Extended Treatment OL): Upadacitinib 30 mg From Part 2 OL Upadacitinib 45 mg (Experimental): Participants received upadacitinib 30 mg tablets, orally, QD for 12 weeks (until Week 24) during the ET Period. Participants who received OL upadacitinib 45 mg during Part 2 and did not achieve clinical response at Week 12 were included in this group.
  Interventions: Drug: Upadacitinib

INTERVENTIONS:
Drug: Matching Placebo for Upadacitinib — Matching placebo tablets
  Arms: Part 1 (Double-blind): Placebo
Drug: Upadacitinib — Upadacitinib tablets
  Other Names: ABT-494; RINVOQ®
  Arms: Part 1 (Double-blind): Upadacitinib 45 mg; Part 2 (Open-label): Upadacitinib 45 mg; Part 3 (Extended Treatment DB): Upadacitinib 30 mg From Part 1 DB Upadacitinib 45 mg; Part 3 (Extended Treatment DB): Upadacitinib 45 mg From Part 1 DB Placebo; Part 3 (Extended Treatment OL): Upadacitinib 30 mg From Part 2 OL Upadacitinib 45 mg

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of upadacitinib compared to placebo as induction therapy in participants with moderately and severely active Crohn's disease (CD).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of CD for at least 3 months prior to Baseline.
* Confirmed diagnosis of moderate to severe CD as assessed by stool frequency (SF), abdominal pain (AP) score.
* Evidence of mucosal inflammation based on the Simplified Endoscopic Score for Crohn's disease (SES-CD) on an endoscopy confirmed by a central reader.
* Demonstrated an inadequate response or intolerance to any biologic therapy for infliximab, adalimumab, certolizumab pegol, vedolizumab, and ustekinumab.
* If female, participant must meet the contraception recommendations.

Exclusion Criteria:

* Participant with a current diagnosis of ulcerative colitis or indeterminate colitis.
* Participant not on stable doses of CD related antibiotics, oral aminosalicylates, corticosteroids or methotrexate (MTX).
* Participant with the following ongoing known complications of CD: abscess (abdominal or peri-anal), symptomatic bowel strictures, fulminant colitis, toxic megacolon, or any other manifestation that might require surgery while enrolled in the study.
* Participant with ostomy or ileoanal pouch.
* Participant diagnosed with conditions that could interfere with drug absorption including but not limited to short gut or short bowel syndrome.
* Screening laboratory and other protocol pre-specified analyses show abnormal results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 624 (Actual)
Dates: Start 2017-11-29 (Actual); Primary Completion 2021-08-11 (Actual); Study Completion 2021-08-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (428):
- United States (119):
  - East View Medical Research, LLC /ID# 171133, Mobile, Alabama
  - CB Flock Research Corporation /ID# 166220, Mobile, Alabama
  - Delsol Research Management, Ll /Id# 170179, Chandler, Arizona
  - HonorHealth Research Institute - Shea /ID# 164734, Scottsdale, Arizona
  - Arizona Arthritis & Rheumatology Research, PLLC /ID# 203891, Sun City, Arizona
  - Southern California Res. Ctr. /ID# 169654, Coronado, California
  - Citrus Valley Gastroenterology /ID# 166201, Covina, California
  - United Medical Doctors /ID# 207452, Los Alamitos, California
  - Gastrointestinal Biosciences Clinical Trials, LLC /ID# 164887, Los Angeles, California
  - Facey Medical Foundation /ID# 203137, Mission Hills, California
  - United Medical Doctors - Murrieta /ID# 164845, Murrieta, California
  - Ucsd /Id# 164679, San Diego, California
  - Medical Assoc Research Grp /ID# 169705, San Diego, California
  - UCSF Center for Colitis and Crohn's Disease /ID# 202373, San Francisco, California
  - Univ of California San Francis /ID# 164843, San Francisco, California
  - Care Access Research /ID# 167766, San Pablo, California
  - Peak Gastroenterology Associates, PC /ID# 170181, Colorado Springs, Colorado
  - Delta Waves, Inc. /ID# 164872, Colorado Springs, Colorado
  - Duplicate_Western States Clinical Research, Inc. /ID# 164895, Wheat Ridge, Colorado
  - Medical Research Center of CT /ID# 164829, Hamden, Connecticut
  - Clinical Research of West Florida, Inc /ID# 205825, Clearwater, Florida
  - Clinical Research of West Florida, Inc /ID# 208117, Clearwater, Florida
  - Advanced Research - Coral Springs /ID# 218020, Coral Springs, Florida
  - Encore Borland-Groover Clinical Research /Id# 203498, Jacksonville, Florida
  - Ctr for Advanced Gastroenterol /ID# 165332, Maitland, Florida
  - Crystal Pharmacology Research /ID# 166101, Miami, Florida
  - Coral Research Clinic /ID# 164657, Miami, Florida
  - Advanced Research Institute, Inc /ID# 164814, New Port Richey, Florida
  - Endoscopic Research, Inc. /ID# 205893, Orlando, Florida
  - Omega Research Maitland, LLC /ID# 203480, Orlando, Florida
  - Clinical Research Trials of Florida, Inc. /ID# 203484, Tampa, Florida
  - AdventHealth Tampa /ID# 171175, Tampa, Florida
  - Gastroenterology Associates of Central Georgia, LLC /ID# 165460, Macon, Georgia
  - Gastroenterology Consultants PC - Roswell /ID# 218219, Roswell, Georgia
  - Atlanta Gastroenterology Spec /ID# 164780, Suwanee, Georgia
  - University of Chicago Medicine /ID# 165472, Chicago, Illinois
  - DuPage Medical Group /ID# 205303, Downers Grove, Illinois
  - MediSphere Medical Research Center /ID# 166209, Evansville, Indiana
  - Indianapolis Gastroenterology /ID# 164837, Indianapolis, Indiana
  - Aquiant Research /ID# 205504, New Albany, Indiana
  - University of Iowa Hospitals and Clinics /ID# 165330, Iowa City, Iowa
  - Tri-State Gastroenterology /ID# 165484, Crestview Hills, Kentucky
  - University of Louisville /ID# 168536, Louisville, Kentucky
  - University of Louisville /ID# 208093, Louisville, Kentucky
  - CroNOLA, LLC /ID# 164722, Houma, Louisiana
  - Nola Research Works, LLC /ID# 164897, New Orleans, Louisiana
  - Louisana Research Center, LLC /ID# 164659, Shreveport, Louisiana
  - Johns Hopkins University School of Medicine /ID# 211940, Baltimore, Maryland
  - MGG Group Co, Inc.Chevy Chase Clinical Research /ID# 164835, Chevy Chase, Maryland
  - Gastro Center of Maryland /ID# 171171, Columbia, Maryland
  - Lahey Hospital and Medical Center /ID# 214725, Burlington, Massachusetts
  - University of Michigan Health Systems /ID# 164844, Ann Arbor, Michigan
  - Clin Res Inst of Michigan, LLC /ID# 170178, Chesterfield, Michigan
  - Digestive Health Associates (DHA) - Farmington Hills /ID# 206099, Farmington Hills, Michigan
  - Center for Digestive Health /ID# 164733, Troy, Michigan
  - Mayo Clinic - Rochester /ID# 164868, Rochester, Minnesota
  - Southern Therapy and Advanced Research (STAR) LLC /ID# 165318, Jackson, Mississippi
  - Quality Clinical Research Inc. /ID# 170177, Omaha, Nebraska
  - CHI Health Research Center /ID# 168545, Omaha, Nebraska
  - Las Vegas Medical Research /ID# 168562, Las Vegas, Nevada
  - AGA Clinical Research Associates, LLC /ID# 164883, Egg Harbor, New Jersey
  - Rutgers Robert Wood Johnson /ID# 166092, New Brunswick, New Jersey
  - NY Scientific /ID# 164833, Brooklyn, New York
  - NYU Langone Long Island Clinical Research Associates /ID# 164830, Lake Success, New York
  - The Mount Sinai Hospital /ID# 170172, New York, New York
  - Columbia Univ Medical Center /ID# 164870, New York, New York
  - Gastro Group of Rochester /ID# 166216, Rochester, New York
  - Richmond University Medical Center /ID# 201855, Staten Island, New York
  - Montefiore Medical Center - Moses Campus /ID# 166226, The Bronx, New York
  - Advantage Clinical Trials /ID# 168557, The Bronx, New York
  - Atrium Health Carolinas Medical Center /ID# 164834, Charlotte, North Carolina
  - PMG Research of Charlotte /ID# 171170, Charlotte, North Carolina
  - Wake Radiology UNC REX Healthcare - Raleigh Office /ID# 164663, Raleigh, North Carolina
  - Wake Forest Baptist Medical Center /ID# 201225, Winston-Salem, North Carolina
  - Plains Clinical Research Center, LLC /ID# 170184, Fargo, North Dakota
  - Consultants for Clinical Research /ID# 164855, Cincinnati, Ohio
  - University of Cincinnati /ID# 164720, Cincinnati, Ohio
  - Cleveland Clinic Main Campus /ID# 208220, Cleveland, Ohio
  - The Ohio State University /ID# 170174, Columbus, Ohio
  - Optimed Research, Ltd. /ID# 205618, Columbus, Ohio
  - Hometown Urgent Care and Resea /ID# 201290, Dayton, Ohio
  - Dayton Gastroenterology, Inc. /ID# 167624, Englewood, Ohio
  - Great Lakes Medical Research, LLC /ID# 202007, Mentor, Ohio
  - Digestive Disease Specialists /ID# 201062, Oklahoma City, Oklahoma
  - Options Health Research, LLC /ID# 164737, Tulsa, Oklahoma
  - Healthcare Research Consultant /ID# 166228, Tulsa, Oklahoma
  - University of Pennsylvania /ID# 168402, Philadelphia, Pennsylvania
  - Thomas Jefferson University /ID# 168014, Philadelphia, Pennsylvania
  - Pharmacorp Clinical Trials /ID# 164809, Charleston, South Carolina
  - Gastroenterology Associates, P.A. of Greenville /ID# 164880, Greenville, South Carolina
  - Rapid City Medical Center - GI Research /ID# 201734, Rapid City, South Dakota
  - Gastro One /ID# 164718, Germantown, Tennessee
  - East Tennessee Research Institute /ID# 203612, Johnson City, Tennessee
  - Quality Medical Research /ID# 205262, Nashville, Tennessee
  - Vanderbilt University Medical Center /ID# 164846, Nashville, Tennessee
  - TX Clinical Research Institute /ID# 164848, Arlington, Texas
  - Inquest Clinical Research /ID# 164865, Baytown, Texas
  - Texas Digestive Disease Consultants /ID# 209952, Cedar Park, Texas
  - Texas Digestive Disease Consultants /ID# 209802, Cedar Park, Texas
  - CliniCore International, LLC /ID# 164662, Houston, Texas
  - Baylor College of Medicine - Baylor Medical Center /ID# 164847, Houston, Texas
  - Centex Studies, Inc. - Houston /ID# 201213, Houston, Texas
  - GI Specialists of Houston /ID# 202338, Houston, Texas
  - Caprock Gastro Research /ID# 215437, Lubbock, Texas
  - Clinical Associates in Research Therapeutics of America, LLC /ID# 164863, San Antonio, Texas
  - Southern Star Research Institute, LLC /ID# 169754, San Antonio, Texas
  - Carl R. Meisner Medical Clinic /ID# 201060, Sugar Land, Texas
  - Tyler Research Institute, LLC /ID# 168681, Tyler, Texas
  - Gastro Health & Nutrition - Victoria /ID# 167813, Victoria, Texas
  - HP Clinical Research /ID# 164929, Bountiful, Utah
  - Advanced Research Institute /ID# 164866, Ogden, Utah
  - Duplicate_Care Access Research /ID# 164853, Salt Lake City, Utah
  - Velocity Clinical Research - Salt Lake City /ID# 166095, West Jordan, Utah
  - Washington Gastroenterology Associates /ID# 164721, Bellevue, Washington
  - Virginia Mason - Seattle Orthapedics /ID# 164680, Seattle, Washington
  - University of Washington /ID# 164875, Seattle, Washington
  - The Vancouver Clinic, INC. PS /ID# 164811, Vancouver, Washington
  - Froedtert Memorial Lutheran Hospital /ID# 202286, Milwaukee, Wisconsin
  - Allegiance Research Specialists /ID# 165321, Wauwatosa, Wisconsin
- Argentina (6):
  - Cardio Alem /ID# 211284, San Isidro, Buenos Aires
  - Hospital Italiano de Buenos Aires /ID# 215543, Ciudad Autonoma Buenos Aires, Ciuadad Autonoma de Buenos Aires
  - Gedyt /ID# 210019, Ciudad Autonoma de Buenos Aire, Ciuadad Autonoma de Buenos Aires
  - Cemic /Id# 169184, Ciudad Autonoma de Buenos Aire, Ciuadad Autonoma de Buenos Aires
  - Hospital Provincial del Centenario /ID# 171254, Rosario, Santa Fe Province
  - Hospital Privado Univesitario /ID# 169228, Córdoba
- Australia (6):
  - Concord Repatriation General Hospital /ID# 171509, Concord, New South Wales
  - Coral Sea Clinical Research institute /ID# 212987, North Mackay, Queensland
  - Mater Misericordiae Limited /ID# 204908, South Brisbane, Queensland
  - Royal Adelaide Hospital /ID# 171511, Adelaide, South Australia
  - Box Hill Hospital /ID# 203734, Box Hill, Victoria
  - Fiona Stanley Hospital /ID# 171510, Murdoch, Western Australia
- Austria (3):
  - Klinik Landstrasse /ID# 203437, Vienna, Vienna
  - Medizinische Universitaet Wien /ID# 169462, Vienna, Vienna
  - Landeskrankenhaus Salzburg-Universitätsklinikum der PMU (LKH) /ID# 214467, Salzburg
- Belgium (5):
  - UCL Saint-Luc /ID# 200297, Woluwe-Saint-Lambert, Brussels Capital
  - CHU de Liege Sart Tilman /ID# 200299, Liège, Liege
  - CHU UCL Namur - site Godinne /ID# 200300, Godinne, Namur
  - Universitair Ziekenhuis Leuven /ID# 200298, Leuven, Vlaams-Brabant
  - AZ Sint-Lucas /ID# 200301, Ghent
- Bosnia and Herzegovina (4):
  - University Clinical Centre of the Republic of Srpska /ID# 208050, Banja Luka, Republika Srpska
  - University Clinical Center Tuzla /ID# 210324, Tuzla, Tuzlanski
  - Clinical Center University of Sarajevo /ID# 203885, Sarajevo
  - Polyclinic and Daily Hospital Dr. Al-Tawil /ID# 217841, Sarajevo
- Brazil (7):
  - Instituto Goiano de Gastroenterologia e Endoscopia Digestiva /ID# 166870, Goiânia, Goiás
  - Hospital Nossa Senhora das Graças /ID# 166869, Curitiba, Paraná
  - Hospital de Clinicas de Porto Alegre /ID# 166872, Porto Alegre, Rio Grande do Sul
  - Upeclin Fmb - Unesp /Id# 166876, Botucatu, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina de Ribeirao Preto - USP /ID# 166874, Ribeirão Preto, São Paulo
  - Faculdade de Medicina do ABC /ID# 208327, Santo André, São Paulo
  - Kaiser Clinica e Hospital Dia /ID# 166873, São José do Rio Preto, São Paulo
- Bulgaria (3):
  - UMHAT Kaspela EOOD /ID# 167617, Plovdiv
  - Duplicate_Second MHAT Sofia /ID# 167618, Sofia
  - MHAT Trakia /ID# 201678, Stara Zagora
- Canada (15):
  - University of Calgary - Cumming School of Medicine - Adult Cystic Fibrosis Clini /ID# 166963, Calgary, Alberta
  - Allen Whey Khye Lim Professional Corporation /ID# 168041, Edmonton, Alberta
  - Covenant Health /ID# 166966, Edmonton, Alberta
  - Fraser Clinical Trials Inc /ID# 166957, New Westminster, British Columbia
  - GIRI Gastrointestinal Research Institute /ID# 166964, Vancouver, British Columbia
  - QEII - Health Sciences Centre /ID# 169306, Halifax, Nova Scotia
  - Medicor Research Inc /ID# 166967, Greater Sudbury, Ontario
  - Scott Shulman Medicine Professional Corporation /ID# 169064, North Bay, Ontario
  - Taunton Surgical Centre /ID# 168039, Oshawa, Ontario
  - The Ottawa Hospital /ID# 212413, Ottawa, Ontario
  - Toronto Digestive Disease Asso /ID# 166961, Vaughan, Ontario
  - CHAU- Hotel-Dieu de Levis /ID# 166958, Lévis, Quebec
  - Crchum /Id# 170121, Montreal, Quebec
  - Montreal General Hospital - McGill University Health Center /ID# 170010, Montreal, Quebec
  - CIUSSS de l'Estrie - CHUS /ID# 170935, Sherbrooke, Quebec
- Chile (5):
  - M y F Estudios Clínicos /ID# 169995, Santiago, Region Metropolitana Santiago
  - Research Group /ID# 203180, Santiago, Santiago Metropolitan
  - Hospital Guillermo Grant Benavente de Concepción /ID# 212422, Concepción
  - CTR Estudios Clinicos /ID# 200650, Providencia
  - Hospital Clinico Universidad De Los Andes /ID# 207465, Santiago
- China (15):
  - Zhongshan Hospital Xiamen University /ID# 204985, Fujian, Anhui
  - Sun Yat-sen Memorial Hospital of Sun Yat-sen University /ID# 205226, Guangzhou, Guangdong
  - The Sixth Affiliated Hosp Sun /ID# 204049, Guangzhou, Guangdong
  - Union Hospital Tongji Medical College Huazhong University of Science and Technol /ID# 204096, Wuhan, Hubei
  - Nanjing Drum Tower Hospital /ID# 204869, Nanjing, Jiangsu
  - The First Affiliated Hospital of Nanchang University /ID# 204070, Nanchang, Jiangxi
  - The First Hospital of Jilin University /ID# 206867, Changchun, Jilin
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine /ID# 204072, Shanghai, Shanghai Municipality
  - The second Affiliated hospital of Zhejiang University school of Medicine /ID# 204078, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital,Meical School Zhejiang University /ID# 204068, Hangzhou, Zhejiang
  - Beijing Friendship Hospital /ID# 204536, Beijing
  - The Second Hospital Central South University /ID# 204075, Changsha
  - Nanfang Hospital of Southern Medical University /ID# 204074, Guangzhou
  - Duplicate_Tianjin Med Univ General Hosp /ID# 206993, Tianjin
  - Tongji Hospital Tongji Medical College Huazhong University of Science and Techno /ID# 204069, Wuhan
- Colombia (2):
  - Hospital Pablo Tobon Uribe /ID# 202405, Medellín, Antioquia
  - Hospital San Vicente de Paul /ID# 200028, Medellín, Antioquia
- Croatia (6):
  - Clinical Hospital Dubrava /ID# 171186, Zagreb, City of Zagreb
  - Klinicki bolnicki centar Sestre milosrdnice /ID# 171190, Zagreb, City of Zagreb
  - Klinicki bolnicki centar Zagreb /ID# 171201, Zagreb, City of Zagreb
  - Poliklinika Solmed /ID# 211518, Zagreb, City of Zagreb
  - UHC Split /ID# 171206, Split
  - Zadar General Hospital /ID# 205534, Zadar
- Czechia (3):
  - Hepato-Gastroenterologie HK, s.r.o. /ID# 171566, Hradec Králové
  - ResTrial s.r.o. /ID# 208652, Prague
  - ARTROSCAN s.r.o. /ID# 171592, Třebovice
- Denmark (4):
  - Nordsjaellands Hospital /ID# 200613, Frederikssund, Capital Region
  - Herlev Hospital /ID# 200782, Herlev, Capital Region
  - Kobenhavns Universitet - Hvidovre Hospital (HH) /ID# 200611, Hvidovre, Capital Region
  - Duplicate_Sjaellands Universitets Hospital /ID# 200783, Roskilde, Region Sjælland
- Egypt (6):
  - Clinical Research Center, Faculty of Medicine, Alexandria university. /ID# 171010, Alexandria
  - Clinical Research Center, Faculty of Medicine, Alexandria university. /ID# 171015, Alexandria
  - Clinical Research Center, Faculty of Medicine, Cairo university /ID# 209557, Cairo
  - National Hepatology and Tropical Medicine Research Institute /ID# 170990, Cairo
  - Faculty of Medicine Ain Shams Research Institute- Clinical Research Centre /ID# 209565, Cairo
  - Air Force Specialized Hospital /ID# 170995, Cairo
- Tartu University Hospital /ID# 203140, Tartu, Tartu, Estonia
- France (13):
  - Chu de Nice-Hopital L'Archet Ii /Id# 171009, Nice, Alpes-Maritimes
  - HCL - Hôpital Lyon Sud /ID# 171014, Pierre-Bénite, Auvergne-Rhône-Alpes
  - CHU Bordeaux - Hopital Haut Lévêque /ID# 207414, Pessac, Gironde
  - CHRU Lille - Hopital Claude Huriez /ID# 206539, Lille, Hauts-de-France
  - Duplicate_Hopital Saint Eloi /ID# 170646, Montpellier, Herault
  - CHRU Nancy - Hôpitaux de Brabois /ID# 170985, Vandœuvre-lès-Nancy, Meurthe-et-Moselle
  - CHU de SAINT ETIENNE - Hopital Nord /ID# 171018, Saint Priest EN Jarez, Pays de la Loire Region
  - CHU Amiens-Picardie Site Sud /ID# 171016, Amiens, Somme
  - CHRU Tours - Hopital Trousseau /ID# 169786, Chambray-lès-Tours
  - Duplicate_CHU Henri Mondor /ID# 169787, Créteil
  - Polyclinique Grand Sud /ID# 170649, Nîmes
  - CHU Toulouse - Hopital Rangueil /ID# 169785, Toulouse
  - Hopital Beaujon /ID# 171011, Clichy, Île-de-France Region
- Germany (12):
  - Universitatsklinikum Mannheim /ID# 168778, Mannheim, Baden-Wurttemberg
  - Universitaetsklinikum Ulm /ID# 203563, Ulm, Baden-Wurttemberg
  - Universitaetsklinikum Erlangen /ID# 203551, Erlangen, Bavaria
  - Universitaetsklinikum Frankfurt /ID# 203565, Frankfurt am Main, Hesse
  - Zentrum für Gastroenterologie Saar MVZ GmbH /ID# 206740, Saarbrücken, Saarland
  - Universitaetsklinikum Schleswig-Holstein Campus Kiel /ID# 168779, Kiel, Schleswig-Holstein
  - Charite Universitaetsklinikum Berlin - Campus Benjamin Franklin /ID# 169067, Berlin
  - Gastroenterologie am Mexikoplatz /ID# 203573, Berlin
  - Universitaetsmedizin Essen St. Josef Krankenhaus Werden /ID# 203571, Essen
  - Agaplesion Markus Krankenhaus /ID# 168777, Frankfurt am Main
  - Universitaetsklinikum Halle (Saale) /ID# 207454, Halle
  - Medizinisches Versorgungszentrum Portal 10 /ID# 200213, Münster
- Greece (6):
  - General Hospital of Athens Ippokratio /ID# 167036, Athens, Attica
  - General Hospital of Chest Diseases of Athens SOTIRIA /ID# 202103, Athens, Attica
  - Tzaneio general hospital of Piraeus /ID# 206432, Piraeus, Attica
  - University General Hospital of Heraklion PA.G.N.I /ID# 167035, Heraklion, Crete
  - General Hospital of Athens Evaggelismos and Ophthalmiatrio of Athens Polyclinic /ID# 167037, Athens
  - Genl Hosp Thess Ippokrateio /ID# 208824, Thessaloniki
- Queen Mary Hospital /ID# 171217, Hong Kong, Hong Kong
- Hungary (6):
  - CRU Hungary Egeszsegugyi és Szolgaltato Kft. /ID# 205546, Miskolc, Borsod-Abauj Zemplen county
  - Bugat Pal Korhaz /ID# 201889, Gyöngyös, Heves County
  - Obudai Egeszsegugyi Centrum Kft. /ID# 201891, Budapest, Pest County
  - Magyar Honvedseg Egeszsegugyi Kozpont /ID# 201719, Budapest
  - Debreceni Egyetem Kenezy Gyula Egyetemi Korhaz /ID# 201720, Debrecen
  - Mentahaz Maganorvosi Kozpont /ID# 201890, Székesfehérvár
- Mercy University Hospital /ID# 206510, Cork, Ireland
- Israel (7):
  - Soroka University Medical Center /ID# 169912, Beersheba, Southern District
  - Tel Aviv Sourasky Medical Center /ID# 204876, Tel Aviv, Tel Aviv
  - Barzilai Medical Center /ID# 223372, Ashkelon
  - Assaf Harofeh Medical Center /ID# 204870, Be’er Ya‘aqov
  - Hadassah Medical Center-Hebrew University /ID# 169927, Jerusalem
  - Rabin Medical Center /ID# 202635, Petah Tikva
  - Kaplan Medical Center /ID# 170277, Rehovot
- Italy (14):
  - University of Catanzaro /ID# 201920, Catanzaro, Calabria
  - Policlinico Universitario Campus Bio-Medico /ID# 168169, Rome, Lazio
  - Azienda Ospedaliera San Camillo Forlanini /ID# 168170, Rome, Lazio
  - Istituto Clinico Humanitas /ID# 168171, Rozzano, Milano
  - Fondazione PTV Policlinico Tor Vergata /ID# 168174, Rome, Roma
  - Presidio Columbus-Fondazione Policlinico Universitario Agostino Gemelli IRCCS-Un /ID# 168168, Rome, Roma
  - IRCCS Ospedale Sacro Cuore Don Calabria /ID# 168172, Negrar, Verona
  - A.O.U. di Bologna Policlinico S.Orsola-Malpighi /ID# 168173, Bologna
  - A.O. Per L'Emergenza Cannizzaro /ID# 168176, Catania
  - Policlinico San Martino/Univer /ID# 168177, Genova
  - ASST Fatebenefratelli Sacco - Ospedale Fatebenefratelli e Oftalmico /ID# 168167, Milan
  - Azienda Ospedaliero-Universitaria di Modena /ID# 200008, Modena
  - A.O. Ospedali Riuniti Villa Sofia - Cervello /ID# 168175, Palermo
  - Azienda Ospedaliero Universitaria Pisana-Stabilimento di Cisanello /ID# 202420, Pisa
- Japan (46):
  - Aichi Medical University Hospital /ID# 165957, Nagakute-shi, Aichi-ken
  - Nagoya University Hospital /ID# 165955, Nagoya, Aichi-ken
  - Nagoya City University Hospital /ID# 165956, Nagoya, Aichi-ken
  - Toyohashi Municipal Hospital /ID# 200174, Toyohashi, Aichi-ken
  - Hirosaki National Hospital /ID# 165944, Hirosaki-shi, Aomori
  - Toho University Sakura Medical Center /ID# 165949, Sakura-shi, Chiba
  - Kurume University Hospital /ID# 166004, Kurume-shi, Fukuoka
  - National Hospital Organization Takasaki General Medical Center /ID# 167136, Takasaki-shi, Gunma
  - NHO Fukuyama Medical Center /ID# 167139, Fukuyama-shi, Hiroshima
  - Hiroshima University Hospital /ID# 166006, Hiroshima, Hiroshima
  - Asahikawa Medical University Hospital /ID# 167133, Asahikawa-shi, Hokkaido
  - Hokkaido P.W.F.A.C. Sapporo-Kosei General Hospital /ID# 165943, Sapporo, Hokkaido
  - Sapporo Medical University Hospital /ID# 167137, Sapporo, Hokkaido
  - Aoyama Clinic /ID# 166001, Kobe, Hyōgo
  - Hyogo College of Medicine College Hospital /Id# 200173, Nishinomiya-shi, Hyōgo
  - Kanazawa University Hospital /ID# 169215, Kanazawa, Ishikawa-ken
  - Iwate Medical University Uchimaru Medical Center /ID# 202407, Morioka, Iwate
  - Imamura General Hospital /ID# 227136, Kagoshima, Kagoshima-ken
  - Idzuro Imamura Hospital /ID# 206651, Kagoshima, Kagoshima-ken
  - Sameshima Hospital /ID# 206674, Kagoshima, Kagoshima-ken
  - Japanese Red Cross Kyoto Daiichi Hosital /ID# 165958, Kyoto, Kyoto
  - Kyoto University Hospital /ID# 169888, Kyoto, Kyoto
  - Yokkaichi Hazu Medical Center /ID# 167191, Yokkaichi-shi, Mie-ken
  - Tohoku University Hospital /ID# 167135, Sendai, Miyagi
  - Nara Medical University Hospital /ID# 169216, Kashihara-shi, Nara
  - Kenseikai Dongo Hospital /ID# 208103, Yamatotakada-shi, Nara
  - Niigata University Medical & Dental Hospital /ID# 170044, Niigata, Niigata
  - Ishida Clinic of IBD and Gastroenterology /ID# 167134, Ōita, Oita Prefecture
  - Chikuba Hospital for Proctological and Gastrointestinal Diseases /ID# 166002, Kurashiki-shi, Okayama-ken
  - Okayama University Hospital /ID# 167355, Okayama, Okayama-ken
  - Kinshukai Infusion Clinic /ID# 218871, Osaka, Osaka
  - Osaka City University Hospital /ID# 166007, Osaka, Osaka
  - Osaka University Hospital /ID# 169662, Suita-shi, Osaka
  - Osaka Medical and Pharmaceutical University Hospital /ID# 206324, Takatsuki-shi, Osaka
  - Tokitokai Tokito clinic /ID# 165945, Saitama-shi, Saitama
  - Shiga University of Medical Science Hospital /ID# 167141, Ōtsu, Shiga
  - NHO Shizuoka Medical Center /ID# 167138, Sunto-gun, Shizuoka
  - Tokyo Medical And Dental University, Medical Hospital /ID# 165948, Bunkyo-ku, Tokyo
  - Duplicate_Tokai University Hachioji Hospital /ID# 165951, Hachioji-shi, Tokyo
  - The Jikei University Hospital /ID# 167142, Minato-ku, Tokyo
  - Kyorin University Hospital /ID# 165950, Mitaka-shi, Tokyo
  - Tokyo Women's Medical University Hospital /ID# 205981, Shinjuku-ku, Tokyo
  - Toyama Prefectural Central Hospital /ID# 217833, Toyama, Toyama
  - Japanese Red Cross Wakayama Medical Center /ID# 200638, Wakayama, Wakayama
  - Wakayama Medical University Hospital /ID# 169481, Wakayama, Wakayama
  - Yamagata University Hospital /ID# 200156, Yamagata, Yamagata
- Latvia (3):
  - Pauls Stradins Clinical University Hospital /ID# 169493, Riga
  - Digestive Disease Center Gastro /ID# 169517, Riga
  - Riga East Clinical University Hospital /ID# 169496, Riga
- Lithuania (2):
  - Hospital of Lithuanian University of Health Sciences Kaunas Clinics /ID# 207263, Kaunas
  - Vilnius University Hospital Santaros Klinikos /ID# 203285, Vilnius
- Malaysia (2):
  - Hospital Sultanah Bahiyah /ID# 202627, Alor Star, Kedah
  - Universiti Kebangsaan Malaysia (UKM) Medical Centre /ID# 170778, Kuala Lumpur, Selangor
- Mexico (3):
  - Instituto de Investigaciones Aplicadas a la Neurociencias A.C. /ID# 207143, Durango, Durango
  - Morales Vargas Centro de Investigacion S.C. /ID# 203495, León, Guanajuato
  - Clinica de Investigacion en Reumatologia y Obesidad S.C. /ID# 206779, Guadalajara, Jalisco
- Netherlands (4):
  - Radboud Universitair Medisch Centrum /ID# 166925, Nijmegen, Gelderland
  - Zuyderland Medisch Centrum /ID# 169698, Heerlen, Limburg
  - Academisch Medisch Centrum /ID# 166924, Amsterdam
  - Medisch Spectrum Twente /ID# 170297, Enschede
- Poland (5):
  - Malopolskie Centrum Kliniczne /ID# 202166, Krakow, Lesser Poland Voivodeship
  - Vistamed /ID# 208570, Wroclaw, Lower Silesian Voivodeship
  - Centrum Zdrowia MDM /ID# 200486, Warsaw, Masovian Voivodeship
  - WIP Warsaw IBD Point Profesor Kierkus /ID# 224300, Warsaw, Masovian Voivodeship
  - Centrum Medyczne Reuma Park w Warszawie /ID# 200488, Warsaw, Masovian Voivodeship
- Portugal (5):
  - Hospital da Senhora da Oliveira Guimaraes, EPE /ID# 170225, Guimarães, Braga District
  - Hospital Egas Moniz /ID# 170249, Lisbon, Porto District
  - Unidade Local de Saúde do Alto Minho, EPE - Hospital Conde de Bertiandos /ID# 200606, Ponte de Lima, Viana do Castelo District
  - Hospital Garcia de Orta, EPE /ID# 170234, Almada
  - Centro Hospitalar Universitario de Sao Joao, EPE /ID# 170231, Porto
- Puerto Rico (2):
  - Mindful Medical Research /ID# 203357, San Juan
  - School of Medicine University of Puerto Rico-Medical Science Campus /ID# 166770, San Juan
- Romania (3):
  - Institutul Clinic Fundeni /ID# 167826, Sector 2, București
  - Clinica GASTRO MED SRL /ID# 206367, Cluj-Napoca, Cluj
  - Cabinet Particular Policlinic Algomed /ID# 167827, Timișoara
- Russia (12):
  - Immanuel Kant Baltic Federal University /ID# 202128, Kaliningrad, Kaliningrad Oblast
  - LLC Medical Center /ID# 209233, Novosibirsk, Novosibirsk Oblast
  - Perm Clinical Center of the Federal Medical and Biological Agency /ID# 202988, Perm, Permskiy Kray
  - LLC Novaya Klinika /ID# 206615, Pyatigorsk, Stavropol Kray
  - Professor Pasechnikov Gastroenterology and Pankreatology clinic /ID# 202995, Stavropol, Stavropol Kray
  - Kazan State Medical University /ID# 169574, Kazan', Tatarstan, Respublika
  - Olla-Med Clinic /ID# 208721, Moscow
  - P.A. Bayandin Murmansk Regiona /ID# 169575, Murmansk
  - Republican hospital named after V.A. Baranov /ID# 206487, Petrozavodsk
  - Euromedservice /ID# 206609, Pushkin
  - X7 Clinical Research Center /ID# 216349, Saint Petersburg
  - City Clinical Hospital No. 31 /ID# 208870, Saint Petersburg
- Serbia (6):
  - Clinical Hosp Center Zvezdara /ID# 168221, Belgrade, Beograd
  - Military Medical Academy /ID# 168784, Belgrade, Beograd
  - University Clinical Center Serbia /ID# 168220, Belgrade, Beograd
  - Clin Hosp Ctr Bezanijska Kosa /ID# 168799, Belgrade, Beograd
  - University Clinical Center Kragujevac /ID# 205858, Kragujevac, Sumadijski Okrug
  - Clinical Center Vojvodina /ID# 168222, Novi Sad, Vojvodina
- Singapore (3):
  - KL Ling Gastroenterology and Liver Clinic /ID# 217963, Singapore
  - Gleneagles Medical Centre /ID# 206530, Singapore
  - Tan Tock Seng Hospital /ID# 203159, Singapore
- Slovakia (2):
  - Fakultna nemocnica s poliklinikou F.D. Roosevelta Banska Bystrica /ID# 169952, Banská Bystrica
  - KM Management, spol. s.r.o. /ID# 170199, Nitra
- Univ Medical Ctr Ljubljana /ID# 211042, Ljubljana, Slovenia
- South Africa (5):
  - Farmovs (Pty) Ltd /Id# 207536, Bloemfontein, Free State
  - Lenasia Clinical Trial Centre /ID# 205144, Johannesburg, Gauteng
  - Wits Clinical Research Site /ID# 170851, Johannesburg, Gauteng
  - Dr JP Wright /ID# 170885, Cape Town, Western Cape
  - Private Practice Dr MN Rajabally /ID# 169852, Cape Town, Western Cape
- South Korea (10):
  - Hayang University GuriHospital /ID# 167578, Guri-si, Gyeonggido
  - CHA University Bundang Medical Center /ID# 167583, Seongnam-si, Gyeonggido
  - Kangbuk Samsung Hospital /ID# 167577, Seoul, Seoul Teugbyeolsi
  - Yonsei University Health System Severance Hospital /ID# 167581, Seoul, Seoul Teugbyeolsi
  - Inje University Haeundae Hospital /ID# 202629, Busan
  - Dong-A University Hospital /ID# 167582, Busan
  - Pusan National University Hospital /ID# 167580, Busan
  - Kyungpook National Univ Hosp /ID# 207015, Daegu
  - Samsung Medical Center /ID# 167579, Seoul
  - Chung-Ang University Hostipal /ID# 207017, Seoul
- Spain (12):
  - Hospital Universitari Son Espases /ID# 201997, Palma de Mallorca, Balearic Islands
  - Hospital Unversitario Marques de Valdecilla /ID# 202039, Santander, Cantabria
  - Hospital Universitario Dr. Negrin /ID# 171238, Las Palmas de Gran Canaria, Las Palmas
  - Complejo Hospitalario de Navarra /ID# 202038, Pamplona, Navarre
  - Hospital Universitario A Coruna - CHUAC /ID# 203908, A Coruña
  - Hospital Universitario Vall d'Hebron /ID# 171237, Barcelona
  - Hospital Clinic de Barcelona /ID# 171242, Barcelona
  - Hospital Universitario de Girona Doctor Josep Trueta /ID# 202040, Girona
  - Hospital Juan Ramon Jimenez /ID# 171243, Huelva
  - Hospital Universitario La Paz /ID# 171241, Madrid
  - Hospital Universitario Virgen Macarena /ID# 171240, Seville
  - Hospital Universitario y Politecnico La Fe /ID# 201988, Valencia
- Sweden (4):
  - Hallands Hospital Halmstad /ID# 170840, Halmstad, Halland County
  - Alingsas lasarett /ID# 170838, Alingsås, Västra Götaland County
  - Sodra Alvsborgs sjukhus /ID# 202889, Borås, Västra Götaland County
  - Sahlgrenska University Hospital /ID# 169031, Gothenburg, Västra Götaland County
- Switzerland (2):
  - Universitätsspital Zürich /ID# 170999, Zurich, Canton of Zurich
  - Inselspital, Universitätsspital Bern /ID# 171006, Bern
- Taiwan (2):
  - National Taiwan University Hospital /ID# 169789, Taipei
  - Linkou Chang Gung Memorial Ho /ID# 169788, Taoyuan
- Turkey (Türkiye) (10):
  - Acibadem Kozyatagi Hospital /ID# 209405, Kadıköy, Istanbul
  - Erciyes University Medical Fac /ID# 171321, Melikgazi, Kayseri
  - Ankara Univ Medical Faculty /ID# 206412, Ankara
  - Inonu Universitesi Turgut Ozal /ID# 201267, Battalgazi/malatya
  - Mustafa Kemal University Medic /ID# 171318, Hatay
  - Istanbul University-Cerrahpasa, Cerrahpasa Medical Faculty /ID# 200280, Istanbul
  - Marmara Universitesi Pendik Egitim ve Arastirma Hastanesi /ID# 171316, Istanbul
  - Mersin University Medical /ID# 171320, Mersin
  - Sisli Etfal Train & Res Hosp /ID# 171317, Şişli
  - Gazi Universitesi Tip Fakultes /ID# 217443, Yenimahalle
- United Kingdom (14):
  - South Eastern Health and Social Care Trust /ID# 205322, Belfast, Antrim
  - Warrington and Halton Hospitals NHS Foundation Trust /ID# 171388, Warrington, Cheshire West And Chester
  - Warrington and Halton Hospitals NHS Foundation Trust /ID# 209085, Warrington, Cheshire West And Chester
  - Barts Health NHS Trust /ID# 218829, London, London, City of
  - Royal United Hospitals Bath /ID# 169084, Bath
  - University Hospitals Birmingham NHS Foundation Trust /ID# 169080, Birmingham
  - The Dudley Group NHS Foundation Trust /ID# 169079, Dudley
  - London North West University Healthcare NHS Trust /ID# 169078, Harrow
  - King's College Hospital NHS Foundation Trusts /ID# 169082, London
  - The Newcastle Upon Tyne Hospitals NHS Foundation Trust /ID# 169085, Newcastle upon Tyne
  - Stockport NHS foundation trust /ID# 208718, Stockport
  - Taunton and Somerset NHS Foundation Trust /ID# 209664, Taunton
  - St George's University Hospitals NHS Foundation Trust /ID# 205551, Tooting
  - The Royal Wolverhampton NHS Trust /ID# 171387, Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing, please refer to the link below.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Use Agreement (DUA). For more information on the process, or to submit a request, visit the following link.
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Derived] Vermeire S, Colombel JF, Danese S, Panaccione R, Peyrin-Biroulet L, Beck K, Chaparro M, Gisbert JP, Dubcenco E, Klaff J, Naling G, Ford S, Remple V, Joshi N, Suravaram S, Duncan B, Wang Y, Wick-Urban B, Loftus EV. Benefit-risk profile of upadacitinib: exploratory post hoc analysis of phase 2b/3 studies in patients with moderately to severely active ulcerative colitis or Crohn's disease. J Crohns Colitis. 2026 Jan 9;20(1):jjaf198. doi: 10.1093/ecco-jcc/jjaf198. PMID 41264726
- [Derived] Dubinsky MC, D'Haens G, Dewit O, Juillerat P, Panaccione R, Fujii T, Dubcenco E, Lacerda AP, Anyanwu SI, Ford S, Cunneen C, Fish I, Joshi N, Garrison A, Loftus EV. Efficacy and Safety with Upadacitinib by Baseline Corticosteroid Use in Patients with Moderately to Severely Active Crohn's Disease. Inflamm Bowel Dis. 2025 Nov 4:izaf250. doi: 10.1093/ibd/izaf250. Online ahead of print. PMID 41189093
- [Derived] Colombel JF, Lacerda AP, Irving PM, Panaccione R, Reinisch W, Rieder F, Steinlauf A, Schwartz D, Feng T, Dubcenco E, Anyanwu SI, Laroux FS, Cunneen C, Powell N. Efficacy and Safety of Upadacitinib for Perianal Fistulizing Crohn's Disease: A Post Hoc Analysis of 3 Phase 3 Trials. Clin Gastroenterol Hepatol. 2025 May;23(6):1019-1029. doi: 10.1016/j.cgh.2024.08.032. Epub 2024 Sep 24. PMID 39326583
- [Derived] Panes J, Louis E, Bossuyt P, Joshi N, Lee WJ, Lacerda AP, Kligys K, Xuan S, Shukla N, Loftus EV Jr. Induction of Endoscopic Response, Remission, and Ulcer-Free Endoscopy With Upadacitinib Is Associated With Improved Clinical Outcomes and Quality of Life in Patients With Crohn's Disease. Inflamm Bowel Dis. 2025 Feb 6;31(2):394-403. doi: 10.1093/ibd/izae200. PMID 39231444
- [Derived] Peyrin-Biroulet L, Panaccione R, Louis E, Atreya R, Rubin DT, Lindsay JO, Siffledeen J, Lukin DJ, Wright J, Watanabe K, Ford S, Remple VP, Lacerda AP, Dubcenco E, Garrison A, Zhou Q, Berg S, Anyanwu SI, Schreiber S. Upadacitinib Achieves Clinical and Endoscopic Outcomes in Crohn's Disease Regardless of Prior Biologic Exposure. Clin Gastroenterol Hepatol. 2024 Oct;22(10):2096-2106. doi: 10.1016/j.cgh.2024.02.026. Epub 2024 Mar 15. PMID 38492904
- [Derived] Colombel JF, Hisamatsu T, Atreya R, Bresso F, Thin L, Panaccione R, Parra RS, Ford S, Remple VP, Lacerda AP, Anyanwu SI, Mallick M, Garrison A, Regueiro M. Upadacitinib Reduces Crohn's Disease Symptoms Within the First Week of Induction Therapy. Clin Gastroenterol Hepatol. 2024 Aug;22(8):1668-1677. doi: 10.1016/j.cgh.2024.02.027. Epub 2024 Mar 15. PMID 38492903
- [Derived] Loftus EV Jr, Panes J, Lacerda AP, Peyrin-Biroulet L, D'Haens G, Panaccione R, Reinisch W, Louis E, Chen M, Nakase H, Begun J, Boland BS, Phillips C, Mohamed MF, Liu J, Geng Z, Feng T, Dubcenco E, Colombel JF. Upadacitinib Induction and Maintenance Therapy for Crohn's Disease. N Engl J Med. 2023 May 25;388(21):1966-1980. doi: 10.1056/NEJMoa2212728. PMID 37224198
- See also: RINVOQ® (upadacitinib) extended-release tablets prescribing information — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study had 3 Parts:
  Part 1:randomized,double-blind,placebo-controlled InductionPeriod(IP); Part 2:Once enrollment for Part1 completed,participants were further enrolled in open-label,single-arm active IP to receive upadacitinib 45mg.Clinical non-responders from Parts1 and 2 entered Part3; Part 3:ExtendedTreatmentPeriod for non-responders from Part1 or 2 had 3 cohorts:Cohort 1=placebo participants from Part 1,Cohort2=upadacitinib participants from Part 1.Cohort3=participants from Part2.
Period: Period 1: DB and OL Induction (12 Weeks)
Arm/Group | Part 1 (Double-blind): Placebo | Part 1 (Double-blind): Upadacitinib 45 mg | Part 2 (Open-label): Upadacitinib 45 mg | Part 3 (Extended Treatment DB): Upadacitinib 45 mg From Part 1 DB Placebo | Part 3 (Extended Treatment DB): Upadacitinib 30 mg From Part 1 DB Upadacitinib 45 mg | Part 3 (Extended Treatment OL): Upadacitinib 30 mg From Part 2 OL Upadacitinib 45 mg
Started | 171 | 324 | 129 | 0 | 0 | 0
Completed (Completed=completed the study) | 149 | 291 | 123 | 0 | 0 | 0
Not Completed | 22 | 33 | 6 | 0 | 0 | 0
Not completed — Adverse Event | 5 | 17 | 2 | 0 | 0 | 0
Not completed — Withdrew Consent | 8 | 8 | 3 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 8 | 4 | 0 | 0 | 0 | 0
Not completed — Reason not Specified | 1 | 3 | 1 | 0 | 0 | 0
Period: Period 2: 12-Week Extended Treatment
Arm/Group | Part 1 (Double-blind): Placebo | Part 1 (Double-blind): Upadacitinib 45 mg | Part 2 (Open-label): Upadacitinib 45 mg | Part 3 (Extended Treatment DB): Upadacitinib 45 mg From Part 1 DB Placebo | Part 3 (Extended Treatment DB): Upadacitinib 30 mg From Part 1 DB Upadacitinib 45 mg | Part 3 (Extended Treatment OL): Upadacitinib 30 mg From Part 2 OL Upadacitinib 45 mg
Started | 0 | 0 | 0 | 78 | 69 | 14
Completed (Completed=completed the study) | 0 | 0 | 0 | 67 | 51 | 8
Not Completed | 0 | 0 | 0 | 11 | 18 | 6
Not completed — Adverse Event | 0 | 0 | 0 | 8 | 5 | 0
Not completed — Withdrew Consent | 0 | 0 | 0 | 0 | 5 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 2 | 6 | 3
Not completed — Coronavirus Disease (COVID-19) Logistical Restrictions | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Reason not Specified | 0 | 0 | 0 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Population for the 12-week DB Induction Period (Part 1) i.e., ITT1 included all randomized participants who received at least one dose of DB study drug during Part 1. ITT Population for the 12-week OL Induction Period (Part 2) i.e., ITT2 included all participants who received at least one dose of study drug in Part 2.
Groups:
- Part 1 (Double Blind): Placebo: Participants received upadacitinib matching placebo tablets, orally, QD for 12 weeks during the Double-blind Induction Period.
- Part 1 (Double Blind): Upadacitinib 45 mg: Participants received upadacitinib 45 mg tablets, orally, QD for 12 weeks during the Double-blind Induction Period.
- Part 2 (Open Label): Upadacitinib 45 mg: Participants received upadacitinib 45 mg tablets, orally, QD for 12 weeks during the Open-label Induction Period.
- Total: Total of all reporting groups
Arm/Group | Part 1 (Double Blind): Placebo | Part 1 (Double Blind): Upadacitinib 45 mg | Part 2 (Open Label): Upadacitinib 45 mg | Total
Number analyzed (Participants) | 171 | 324 | 129 | 624
Age, Continuous [Mean (Full Range); unit: years] — Population: Results are reported separately for Part 1 (Double Blind) and Part 2 (Open Label.)
  years
    Part 1 (Double Blind): number analyzed (Participants) | 171 | 324 | 0 | 495
    Part 1 (Double Blind) | 37.5 [18 to 74] | 38.4 [18 to 73] |  | 38.1 [18 to 74]
    Part 2 (Open Label): number analyzed (Participants) | 0 | 0 | 129 | 129
    Part 2 (Open Label) |  |  | 39.1 [18 to 68] | 39.1 [18 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 155 | 60 | 290
  Male | 96 | 169 | 69 | 334
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 24 | 8 | 40
  Not Hispanic or Latino | 163 | 300 | 121 | 584
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 2
  Asian | 38 | 69 | 11 | 118
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 6 | 19 | 5 | 30
  White | 126 | 230 | 113 | 469
  More than one race | 0 | 5 | 0 | 5
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Clinical Remission Per Crohn's Disease Activity Index (CDAI) at Week 12
Description: The CDAI was used to evaluate the activity of Crohn's disease. Clinical remission per CDAI is defined as CDAI <150. The CDAI is calculated on the basis of a one-week evaluation of 8 items: frequency of liquid or very soft stool, abdominal pain, complications of Crohn's disease (e.g., uveitis, arthritis, fistula, and abscess), abdominal mass, hematocrit, body weight, use of antidiarrheals, and general condition. Total score ranges from 0 to about 600. Higher CDAI scores indicate more severe disease. CDAI scores below 150 represent remission and scores over 450 represent very severe Crohn's disease. Results were based on non-responder imputation incorporating multiple imputation to handle missing data due to COVID-19 (NRI-C).
Time Frame: Week 12
Population: ITT1 Population included all randomized participants who received at least one dose of DB study drug during Part 1.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Part 1 (Double Blind): Placebo: Participants received upadacitinib matching placebo tablets, orally, QD for 12 weeks during the DB Induction Period.
- Part 1 (Double Blind): Upadacitinib 45 mg: Participants received upadacitinib 45 mg tablets, orally, QD for 12 weeks during the DB Induction Period.
Arm/Group | Part 1 (Double Blind): Placebo | Part 1 (Double Blind): Upadacitinib 45 mg
Number analyzed (Participants) | 171 | 324
percentage of participants | 21.1 [14.9 to 27.2] | 38.9 [33.6 to 44.2]
Statistical Analysis 1: Comparison: Part 1 (Double Blind): Placebo vs Part 1 (Double Blind): Upadacitinib 45 mg; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was calculated using Cochran-Mantel Haenszel (CMH) test adjusted for randomization stratification factors; Adjusted Risk Difference = 17.9, 95% CI 2-sided [10.0 to 25.8] — Point estimate and 95% confidence interval (CI) were calculated using CMH risk difference estimate

2. Primary Outcome: Percentage of Participants With Endoscopic Response at Week 12
Description: Endoscopic response was defined as greater than 50% decrease in Simple Endoscopic Score for Crohn's Disease (SES-CD) from Baseline of the induction study (or for participants with an SES-CD of 4 at Baseline of the induction study, at least a 2-point reduction from Baseline), as scored by Central Reviewer. SES-CD is calculated based on the sum of individual segment values for four endoscopic variables (presence and size of ulcers, ulcerated surface, affected surface and presence of narrowing). Each variable in each segment is scored 0 to 3 resulting in SES-CD values ranging from 0 to 56 with higher scores indicating more severe disease. Results were based on NRI-C.
Time Frame: Baseline to Week 12
Population: ITT1 Population included all randomized participants who received at least one dose of DB study drug during Part 1.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1 (Double Blind): Placebo | Part 1 (Double Blind): Upadacitinib 45 mg
Number analyzed (Participants) | 171 | 324
percentage of participants | 3.5 [0.8 to 6.3] | 34.6 [29.4 to 39.8]
Statistical Analysis 1: Comparison: Part 1 (Double Blind): Placebo vs Part 1 (Double Blind): Upadacitinib 45 mg; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was calculated using CMH test adjusted for randomization stratification factors; Adjusted Risk Difference = 31.2, 95% CI 2-sided [25.5 to 37.0] — Point estimate and 95% CI was calculated using CMH risk difference estimate

3. Primary Outcome: Number of Participants With Adverse Events
Description: An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not the event is considered causally related to the use of the product.
Time Frame: From first dose of study drug until 30 days following last dose of study drug (up to approximately 28 weeks)
Population: Safety Population for Part 1 (SA1)=all participants who received at least one dose of the study drug in Part 1,SA2=all participants who received at least one dose of the study drug in Part 2, and SA3=all participants who received at least one dose of the study drug (upadacitinib 30 mg or upadacitinib 45 mg) in Part 3.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 (Double-blind): Placebo | Part 1 (Double-blind): Upadacitinib 45 mg | Part 2 (Open-label): Upadacitinib 45 mg | Part 3 (Extended Treatment DB): Upadacitinib 45 mg From Part 1 DB Placebo | Part 3 (Extended Treatment DB): Upadacitinib 30 mg From Part 1 DB Upadacitinib 45 mg | Part 3 (Extended Treatment OL): Upadacitinib 30 mg From Part 2 OL Upadacitinib 45 mg
Number analyzed (Participants) | 171 | 324 | 129 | 78 | 69 | 14
Participants | 112 | 221 | 86 | 53 | 45 | 9

4. Secondary Outcome: Percentage of Participants With Clinical Remission Per Patient-Reported Outcomes (PROs) at Week 12
Description: Clinical remission per PROs was defined as average daily very soft or liquid stool frequency (SF) ≤2.8 and average daily abdominal pain (AP) score ≤1.0 and both not greater than Baseline. The number of soft or liquid stools and abdominal pain rated on a scale of 0=none to 3=severe were recorded in an electronic diary. Results were based on NRI-C.
Time Frame: Baseline to Week 12
Population: ITT1 Population included all randomized participants who received at least one dose of DB study drug during Part 1.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1 (Double Blind): Placebo | Part 1 (Double Blind): Upadacitinib 45 mg
Number analyzed (Participants) | 171 | 324
percentage of participants | 14.0 [8.8 to 19.2] | 39.8 [34.5 to 45.1]
Statistical Analysis 1: Comparison: Part 1 (Double Blind): Placebo vs Part 1 (Double Blind): Upadacitinib 45 mg; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was calculated using CMH test adjusted for randomization stratification factors; Adjusted Treatment Difference = 25.9, 95% CI 2-sided [18.7 to 33.1] — Point estimate and 95% CI was calculated using CMH

5. Secondary Outcome: Percentage of Participants With Endoscopic Remission at Week 12
Description: Endoscopic remission was defined per SES-CD. SES-CD ≤4 and at least 2-point reduction from Baseline and no subscore >1 in any individual variable, as scored by Central Reviewer. SES-CD is calculated based on the sum of individual segment values for four endoscopic variables (presence and size of ulcers, ulcerated surface, affected surface and presence of narrowing). Each variable in each segment is scored 0 to 3 resulting in SES-CD values ranging from 0 to 56 with higher scores indicating more severe disease. Results were based on NRI-C.
Time Frame: Baseline to Week 12
Population: ITT1 Population included all randomized participants who received at least one dose of DB study drug during Part 1.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1 (Double Blind): Placebo | Part 1 (Double Blind): Upadacitinib 45 mg
Number analyzed (Participants) | 171 | 324
percentage of participants | 2.3 [0.1 to 4.6] | 19.1 [14.9 to 23.4]
Statistical Analysis 1: Comparison: Part 1 (Double Blind): Placebo vs Part 1 (Double Blind): Upadacitinib 45 mg; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was calculated using CMH test adjusted for randomization stratification factors; Adjusted Treatment Difference = 16.8, 95% CI 2-sided [12.0 to 21.6] — Point estimate and 95% CI was calculated using CMH

6. Secondary Outcome: Percentage of Participants Who Discontinued Corticosteroid Use for Crohn's Disease (CD) and Achieved Clinical Remission Per CDAI at Week 12, in Participants Taking Corticosteroids at Baseline
Description: As prespecified in the protocol, this outcome measure was planned to be assessed in participants taking corticosteroids at Baseline. Clinical remission per CDAI: CDAI <150. The CDAI is used to evaluate the activity of Crohn's disease. The CDAI is calculated on the basis of a one-week evaluation of 8 items: frequency of liquid or very soft stool, abdominal pain, complications of Crohn's disease (e.g., uveitis, arthritis, fistula, and abscess), abdominal mass, hematocrit, body weight, use of antidiarrheals, and general condition. Total score ranges from 0 to about 600. Higher CDAI scores indicate more severe disease. CDAI scores below 150 represent remission and scores over 450 represent very severe Crohn's disease. Results were based on NRI-C.
Time Frame: Week 12
Population: ITT1 Population included all randomized participants who received at least one dose of DB study drug during Part 1. Overall Number of Participants Analyzed are the number of participants taking corticosteroids at Baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1 (Double Blind): Placebo | Part 1 (Double Blind): Upadacitinib 45 mg
Number analyzed (Participants) | 60 | 108
percentage of participants | 11.7 [3.5 to 19.8] | 34.3 [25.3 to 43.2]
Statistical Analysis 1: Comparison: Part 1 (Double Blind): Placebo vs Part 1 (Double Blind): Upadacitinib 45 mg; Test type: Superiority; p = 0.0001, Cochran-Mantel-Haenszel — P-value was calculated using CMH test adjusted for randomization stratification factors; Adjusted Treatment Difference = 22.5, 95% CI 2-sided [11.1 to 34.0] — Point estimate and 95% CI was calculated using CMH

7. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) Total Score at Week 12
Description: The FACIT-F questionnaire was developed to assess fatigue associated with anemia. It consists of 13 fatigue-related questions. The responses to the 13 items on the FACIT-F questionnaire are each measured on a 5-point Likert scale. The responses to the answers are the following: 0= not at all; 1= a little bit; 2= somewhat; 3= quite a bit; 4=very much. Thus, the total score ranges from 0 to 52. High scores represent less fatigue. A positive change from Baseline indicates improvement.
Time Frame: Baseline and Week 12
Population: ITT1 Population included all randomized participants who received at least one dose of DB study drug during Part 1. Overall Number of Participants Analyzed are the number of participants with data available at the given timepoint.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Part 1 (Double Blind): Placebo | Part 1 (Double Blind): Upadacitinib 45 mg
Number analyzed (Participants) | 129 | 278
score on a scale | 3.9 (0.97) | 11.4 (0.69)
Statistical Analysis 1: Comparison: Part 1 (Double Blind): Placebo vs Part 1 (Double Blind): Upadacitinib 45 mg; Test type: Superiority; p < 0.0001, MMRM — P-value was calculated using mixed effect model repeat measurement (MMRM) with Baseline, treatment, visit, treatment by visit interaction and stratification factors in the model; Adjusted Treatment Difference = 7.5, 95% CI 2-sided [5.2 to 9.8] — Point estimate and 95% CI was calculated using MMRM

8. Secondary Outcome: Change From Baseline in Inflammatory Bowel Disease Questionnaire (IBDQ) Total Score at Week 12
Description: The IBDQ is a disease-specific instrument composed of 32 Likert-scaled items. The IBDQ scale contains 4 component subscales: bowel symptoms (10 items), systemic symptoms (5 items), emotional function (12 items), and social function(5 items). Each item is scored on a 7-point scale where: 1=worst to 7= best. The total score ranges from 32 to 224, with higher scores indicating better health-related quality of life. A positive change from Baseline indicates improvement.
Time Frame: Baseline and Week 12
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Part 1 (Double Blind): Placebo | Part 1 (Double Blind): Upadacitinib 45 mg
Number analyzed (Participants) | 130 | 280
score on a scale | 21.6 (3.02) | 46.0 (2.14)
Statistical Analysis 1: Comparison: Part 1 (Double Blind): Placebo vs Part 1 (Double Blind): Upadacitinib 45 mg; Test type: Superiority; p < 0.0001, MMRM — P-value was calculated using MMRM with Baseline, treatment, visit, treatment by visit interaction and stratification factors in the model; Adjusted Treatment Difference = 24.3, 95% CI 2-sided [17.2 to 31.5] — Point estimate and 95% CI was calculated using MMRM

9. Secondary Outcome: Percentage of Participants Achieving Clinical Response 100 (CR-100) at Week 2
Description: CR-100 is defined as a decrease of at least 100 points in CDAI from Baseline at Week 2. The CDAI is used to evaluate the activity of Crohn's disease. The CDAI is calculated on the basis of a one-week evaluation of 8 items: frequency of liquid or very soft stool, abdominal pain, complications of Crohn's disease (e.g., uveitis, arthritis, fistula, and abscess), abdominal mass, hematocrit, body weight, use of antidiarrheals, and general condition. Total score ranges from 0 to about 600. Higher CDAI scores indicate more severe disease. CDAI scores below 150 represent remission and scores over 450 represent very severe Crohn's disease. Results were based on NRI-C.
Time Frame: Baseline to Week 2
Population: ITT1 Population included all randomized participants who received at least one dose of DB study drug during Part 1.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1 (Double Blind): Placebo | Part 1 (Double Blind): Upadacitinib 45 mg
Number analyzed (Participants) | 171 | 324
percentage of participants | 12.4 [7.4 to 17.4] | 33.2 [28.0 to 38.3]
Statistical Analysis 1: Comparison: Part 1 (Double Blind): Placebo vs Part 1 (Double Blind): Upadacitinib 45 mg; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was calculated using CMH test adjusted for randomization stratification factors; Adjusted Treatment Difference = 20.7, 95% CI 2-sided [13.7 to 27.8] — Point estimate and 95% CI was calculated using CMH

10. Secondary Outcome: Percentage of Participants Achieving Clinical Response 100 (CR-100) at Week 12
Description: CR-100 is defined as a decrease of at least 100 points in CDAI from Baseline at Week 12. The CDAI is used to evaluate the activity of Crohn's disease. The CDAI is calculated on the basis of a one-week evaluation of 8 items: frequency of liquid or very soft stool, abdominal pain, complications of Crohn's disease (e.g., uveitis, arthritis, fistula, and abscess), abdominal mass, hematocrit, body weight, use of antidiarrheals, and general condition. Total score ranges from 0 to about 600. Higher CDAI scores indicate more severe disease. CDAI scores below 150 represent remission and scores over 450 represent very severe Crohn's disease. Results were based on NRI-C.
Time Frame: Baseline to Week 12
Population: ITT1 Population included all randomized participants who received at least one dose of DB study drug during Part 1.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1 (Double Blind): Placebo | Part 1 (Double Blind): Upadacitinib 45 mg
Number analyzed (Participants) | 171 | 324
percentage of participants | 27.5 [20.8 to 34.2] | 50.5 [45.1 to 56.0]
Statistical Analysis 1: Comparison: Part 1 (Double Blind): Placebo vs Part 1 (Double Blind): Upadacitinib 45 mg; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was calculated using CMH test adjusted for randomization stratification factors; Adjusted Treatment Difference = 22.8, 95% CI 2-sided [14.4 to 31.2] — Point estimate and 95% CI was calculated using CMH

11. Secondary Outcome: Percentage of Participants With Clinical Remission Per Crohn's Disease Activity Index (CDAI) at Week 4
Description: The CDAI was used to evaluate the activity of Crohn's disease. Clinical remission per CDAI is defined as CDAI <150. The CDAI is calculated on the basis of a one-week evaluation of 8 items: frequency of liquid or very soft stool, abdominal pain, complications of Crohn's disease (e.g., uveitis, arthritis, fistula, and abscess), abdominal mass, hematocrit, body weight, use of antidiarrheals, and general condition. Total score ranges from 0 to 600. Higher CDAI scores indicate more severe disease. CDAI scores below 150 represent remission and scores over 450 represent very severe Crohn's disease. Results were based on NRI-C.
Time Frame: Week 4
Population: ITT1 Population included all randomized participants who received at least one dose of DB study drug during Part 1.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1 (Double Blind): Placebo | Part 1 (Double Blind): Upadacitinib 45 mg
Number analyzed (Participants) | 171 | 324
percentage of participants | 17.7 [11.9 to 23.4] | 29.6 [24.7 to 34.6]
Statistical Analysis 1: Comparison: Part 1 (Double Blind): Placebo vs Part 1 (Double Blind): Upadacitinib 45 mg; Test type: Superiority; p = 0.0013, Cochran-Mantel-Haenszel — P-value was calculated using CMH test adjusted for randomization stratification factors; Adjusted Treatment Difference = 12.1, 95% CI 2-sided [4.7 to 19.5] — Point estimate and 95% CI was calculated using CMH

12. Secondary Outcome: Percentage of Participants With Hospitalizations Due to Crohn's Disease (CD) During Part 1 (12-week Double-blind Induction Period)
Time Frame: Up to Week 12 in Part 1: Double-blind Induction Period
Population: ITT1 Population included all randomized participants who received at least one dose of DB study drug during Part 1.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1 (Double Blind): Placebo | Part 1 (Double Blind): Upadacitinib 45 mg
Number analyzed (Participants) | 171 | 324
percentage of participants | 8.8 [4.5 to 13.0] | 6.2 [3.6 to 8.8]
Statistical Analysis 1: Comparison: Part 1 (Double Blind): Placebo vs Part 1 (Double Blind): Upadacitinib 45 mg; Test type: Superiority; p = 0.2834, Chi-squared — P-value was calculated using Chi-squared test; Treatment Difference = -2.6, 95% CI 2-sided [-7.6 to 2.4] — Point estimate and 95% CI was calculated using Chi-squared test

13. Secondary Outcome: Percentage of Participants With Resolution of Extra-Intestinal Manifestations (EIMs) at Week 12, in Participants With EIMs at Baseline
Description: EIMs are defined as manifestations of Crohn's disease in areas of the body other than the digestive tract, including eyes, skin, joints, mouth, and liver. Results were based on NRI-C.
Time Frame: Week 12
Population: ITT1 Population included all randomized participants who received at least one dose of DB study drug during Part 1. Overall Number of Participants Analyzed are the number of participants with any EIMs at Baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1 (Double Blind): Placebo | Part 1 (Double Blind): Upadacitinib 45 mg
Number analyzed (Participants) | 60 | 131
percentage of participants | 21.7 [11.2 to 32.1] | 32.8 [24.8 to 40.9]
Statistical Analysis 1: Comparison: Part 1 (Double Blind): Placebo vs Part 1 (Double Blind): Upadacitinib 45 mg; Test type: Superiority; p = 0.0833, Cochran-Mantel-Haenszel — P-value was calculated using CMH test adjusted for randomization stratification factors; Adjusted Treatment Difference = 11.5, 95% CI 2-sided [-1.5 to 24.4] — Point estimate and 95% CI was calculated using CMH

ADVERSE EVENTS:
Time Frame: From first dose of study drug until 30 days following last dose of study drug (up to approximately 28 weeks)
Description: Safety Population for Part 1 (SA1)=all participants who received at least one dose of the study drug in Part 1,SA2=all participants who received at least one dose of the study drug in Part 2, and SA3=all participants who received at least one dose of the study drug (upadacitinib 30 mg or upadacitinib 45 mg) in Part 3.
Groups:
- Part 1 (Double-blind): Placebo: Participants received upadacitinib matching placebo tablets, orally, QD for 12 weeks during the DB Induction Period.
- Part 2 (Open Label): Upadacitinib 45 mg: Participants received upadacitinib 45 mg tablets, orally, QD for 12 weeks during the OL Induction Period.
- Part 3 (Extended Treatment DB): Upadacitinib 45 mg From Part 1 DB Placebo; Part 3 (Extended Treatment DB): Upadacitinib 30 mg From Part 1 DB Upadacitinib 45 mg: Participants received upadacitinib 45 mg tablets, orally, QD for 12 weeks (until Week 24) during the Extended Treatment Period. Participants who received placebo in Part 1 and did not achieve clinical response at Week 12 were included in this group.
- Part 3 (Extended Treatment OL): Upadacitinib 30 mg From Part 2 OL Upadacitinib 45 mg: Participants received upadacitinib 30 mg tablets, orally, QD for 12 weeks (until Week 24) during the Extended Treatment Period. Participants who received OL upadacitinib 45 mg during Part 2 and did not achieve clinical response at Week 12 were included in this group.
Arm/Group | Part 1 (Double-blind): Placebo | Part 1 (Double Blind): Upadacitinib 45 mg | Part 2 (Open Label): Upadacitinib 45 mg | Part 3 (Extended Treatment DB): Upadacitinib 45 mg From Part 1 DB Placebo | Part 3 (Extended Treatment DB): Upadacitinib 30 mg From Part 1 DB Upadacitinib 45 mg | Part 3 (Extended Treatment OL): Upadacitinib 30 mg From Part 2 OL Upadacitinib 45 mg
All-Cause Mortality (participants affected / at risk) | 0/171 | 1/324 | 0/129 | 0/78 | 0/69 | 0/14
Serious Adverse Events (participants affected / at risk) | 17/171 | 30/324 | 9/129 | 11/78 | 7/69 | 5/14
Other Adverse Events (participants affected / at risk) | 69/171 | 126/324 | 44/129 | 29/78 | 12/69 | 7/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 (Double-blind): Placebo (N=171) | Part 1 (Double Blind): Upadacitinib 45 mg (N=324) | Part 2 (Open Label): Upadacitinib 45 mg (N=129) | Part 3 (Extended Treatment DB): Upadacitinib 45 mg From Part 1 DB Placebo (N=78) | Part 3 (Extended Treatment DB): Upadacitinib 30 mg From Part 1 DB Upadacitinib 45 mg (N=69) | Part 3 (Extended Treatment OL): Upadacitinib 30 mg From Part 2 OL Upadacitinib 45 mg (N=14)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LEUKOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VERTIGO (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COLITIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CROHN'S DISEASE (Gastrointestinal disorders) | 10 (13) | 7 (7) | 4 (4) | 3 (3) | 4 (5) | 3 (3)
ENTEROCUTANEOUS FISTULA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HAEMATOCHEZIA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HAEMORRHOIDS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ILEAL PERFORATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ILEUS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
INTESTINAL PERFORATION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INTESTINAL STENOSIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PANCREATITIS ACUTE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
PYREXIA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CHOLELITHIASIS (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ABDOMINAL WALL ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
ANAL ABSCESS (Infections and infestations) | 2 (2) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
COLONIC ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CYTOMEGALOVIRUS INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GASTROENTERITIS VIRAL (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PNEUMOCYSTIS JIROVECII PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PYELONEPHRITIS ACUTE (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RETROPERITONEAL ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SEPTIC SHOCK (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
POSTOPERATIVE ILEUS (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GOUT (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
TYPE 1 DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANKYLOSING SPONDYLITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DEPRESSION (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DRUG ABUSE (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DRUG USE DISORDER (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PSYCHOTIC DISORDER (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NEPHROLITHIASIS (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
URETEROLITHIASIS (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FEMALE GENITAL TRACT FISTULA (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
UTERINE POLYP (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANGIOEDEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 (Double-blind): Placebo (N=171) | Part 1 (Double Blind): Upadacitinib 45 mg (N=324) | Part 2 (Open Label): Upadacitinib 45 mg (N=129) | Part 3 (Extended Treatment DB): Upadacitinib 45 mg From Part 1 DB Placebo (N=78) | Part 3 (Extended Treatment DB): Upadacitinib 30 mg From Part 1 DB Upadacitinib 45 mg (N=69) | Part 3 (Extended Treatment OL): Upadacitinib 30 mg From Part 2 OL Upadacitinib 45 mg (N=14)
ANAEMIA (Blood and lymphatic system disorders) | 9 (12) | 16 (17) | 6 (6) | 3 (3) | 1 (1) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 11 (13) | 9 (10) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 1 (1) | 7 (7) | 7 (7) | 1 (1) | 0 (0) | 0 (0)
CROHN'S DISEASE (Gastrointestinal disorders) | 13 (13) | 12 (12) | 5 (5) | 5 (5) | 4 (4) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 8 (9) | 15 (15) | 3 (3) | 3 (3) | 1 (1) | 2 (2)
VOMITING (Gastrointestinal disorders) | 4 (5) | 8 (8) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
PYREXIA (General disorders) | 8 (8) | 13 (13) | 4 (5) | 4 (4) | 1 (1) | 0 (0)
FOLLICULITIS (Infections and infestations) | 1 (1) | 5 (5) | 2 (2) | 5 (5) | 0 (0) | 0 (0)
INFLUENZA (Infections and infestations) | 2 (2) | 9 (10) | 1 (1) | 2 (2) | 3 (3) | 1 (1)
NASOPHARYNGITIS (Infections and infestations) | 5 (5) | 23 (24) | 2 (2) | 3 (4) | 2 (2) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 5 (5) | 17 (18) | 1 (1) | 2 (3) | 2 (2) | 0 (0)
BLOOD PHOSPHORUS DECREASED (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 11 (11) | 7 (7) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 11 (12) | 4 (4) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
FISTULA DISCHARGE (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HEADACHE (Nervous system disorders) | 9 (10) | 20 (24) | 8 (8) | 2 (2) | 0 (0) | 0 (0)
INSOMNIA (Psychiatric disorders) | 2 (2) | 5 (5) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
HAEMATURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ACNE (Skin and subcutaneous tissue disorders) | 4 (4) | 15 (16) | 18 (18) | 5 (5) | 0 (0) | 0 (0)
ALOPECIA (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2021-03-05): https://cdn.clinicaltrials.gov/large-docs/36/NCT03345836/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-15): https://cdn.clinicaltrials.gov/large-docs/36/NCT03345836/SAP_001.pdf